CLINICAL TRIAL: NCT03857945
Title: Effect of Preoperative Mobility Device Training on Postoperative Fall Incidence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ashish Shah, Associate Professor, Foot & Ankle Division, Department of Orthopaedics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300002190-001; 021-13307-E (Other Grant/Funding Number: American Orthopedic Foot and Ankle Society)
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Injury; Muscle, Ankle, and Foot, Multiple
Keywords: preoperative mobility device training
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Working in conjunction with UAB Foot and Ankle Division of the Orthopaedic department, volunteers meeting inclusion criteria will be identified in the outpatient clinic setting. After thorough discussion of risks and benefits, potential volunteers will be consented for participation in the study. The volunteer's demographic data will be obtained including gender, age, and race. The patient will then undergo the "pre-operative mobility device(s) training" during the pre-operative physical therapy visit, if they are randomized to Group 1. Patients in Group 2 will not receive this training. The preoperative training will not incur any additional cost to the patient. Patients in both groups will then undergo standard operative care. During routine 2-week and 6-week follow-up visits, they will be asked questions from a questionnaire that will assess the number and details of any fall(s) they may have experienced.
Masking Description: Masking not feasible for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobility Device Training Group (Active Comparator): Patients receiving preoperative mobility device(s) training before surgery
  Interventions: Other: Preoperative mobility device(s) training
- No Mobility Device Training Group (No Intervention): Patients not receiving preoperative mobility device(s) training before surgery

INTERVENTIONS:
Other: Preoperative mobility device(s) training — Patients in Group 1 (the intervention, that is the mobility device training group group) will receive training on the mobility device(s) with the physical therapy visit during their standard pre-operative care.
  Arms: Mobility Device Training Group

SUMMARY:
The purpose of this study is to determine whether preoperative mobility device training is beneficial in reducing incidence of postoperative falls in patients undergoing elective foot and ankle surgery requiring a postoperative period of no weight-bearing.

DETAILED DESCRIPTION:
Most of the surgeries involving the foot and ankle require non-weight bearing status post operatively. Patients use crutches, walker or knee scooters during that period to avoid weight bearing. However, using any mobility device(s) requires training to avoid falls. Most of the falls happen during early post-operative period after any surgery. The usage of assistive mobility device(s) increases the risk of falls. Some studies have shown physical therapy and training to decrease this risk of falls. Physical training for usage of assistive devices can be done either preoperatively or post operatively. When training is done postoperatively, it may increase the risk of fall due to pain, usage of narcotic drugs, especially in older patients due to lack of muscle power. To prevent these increased risks, the training can be done preoperatively. However, the role of preoperative training regarding usage of assistive devices has not been emphasized in the literature. Hence, the aim of our current study is to evaluate the difference between preoperative training and no training before surgery on the use of mobility device(s).

250 patients will be enrolled in the study. Each participant will be stratified by randomization into either Group 1 or Group 2. Patients in Group 1 will receive training on the mobility device(s) during their standard pre-operative care whereas patients in Group 2 will not receive this training. This training is not a component of routine, standard pre-operative care. Each group will include 125 patients.

Working in conjunction with University of Alabama at Birmingham (UAB) Foot and Ankle Division of the Orthopaedic department, volunteers meeting inclusion criteria will be identified in the outpatient clinic setting. After thorough discussion of risks and benefits, potential volunteers will be consented for participation in the study. The volunteer's demographic data will be obtained including gender, age, and race. The patient will then undergo the "pre-operative mobility device(s) training" during the pre-operative physical therapy visit, if they are randomized to Group 1. Patients in Group 2 will not receive this training. The preoperative training will not incur any additional cost to the patient. Patients in both groups will then undergo standard operative care. During routine 2-week and 6-week follow-up visits, they will be asked questions from a questionnaire that will assess the number and details of any fall(s) they may have experienced.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* undergoing elective unilateral foot/ankle surgery
* requiring a period of post-operative non-weight-bearing or partial-weight-bearing period as advised by the operating surgeon.

Exclusion Criteria:

* less than 18 years of age
* wheelchair-bound patients
* patients with history of previous use of post-operative mobility device(s)
* patients with ankle fractures, patients with previously diagnosed condition(s) with cognitive, balance, mobility impairment
* patients undergoing bilateral surgery
* patients requiring follow ups longer than 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of falls in the post-operative period after foot and ankle surgery | two weeks before surgery to six weeks after surgery
  Number of falls in the post-operative period after foot and ankle surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ashish B Shah, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No